CLINICAL TRIAL: NCT01660490
Title: Development and Validation of Intraoperative Image-quality Criteria A Retrospective Multicenter Case Series to Validate a Set of Intraoperative Image-quality Criteria
Brief Title: Development and Validation of Intraoperative Image-quality Criteria
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: IO Image Quality
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Proximal Femur Fractures
Keywords: Radiographic Image Enhancement,; Intraoperative Care; Femoral Fractures; Femoral Neck Fractures; Hip Fractures, Internal Fixators; Fracture Fixation Internal; Fracture Fixation Intramedullary; Fractures Bone
MeSH Terms: conditions — Proximal Femoral Fractures; Femoral Fractures; Femoral Neck Fractures; Hip Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Proximal femur fractures with ORIF: Proximal femur fractures treated with ORIF
  Interventions: Procedure: ORIF

INTERVENTIONS:
Procedure: ORIF — Open reduction internal fixation of the proximal femur

SUMMARY:
An expert panel of surgeons agreed that there is not any established, standardized approach to the teaching of intraoperative imaging and that there may be practice gaps in decision making and the use of imaging among trauma surgeons.

The panel is set to initiate a consensus-based evaluation process to develop a list of criteria for assessing images and would like to validate these criteria for differentiating good quality versus poor quality images in term of reliability and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of proximal femur fracture
* Operated between May 2010 and December 2010
* Open Reduction Internal Fixation (ORIF)
* Lateral and anteroposterior intraoperative images available

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a proximal femur fractures treated with ORIF between May 2010 and December 2010
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Evaluate if C-Arm pictures can be a predictive factor for the outcome of repositioning of humerus fractures. | Intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blauth, Professor, Principal Investigator — Medical University Innsbruck
Locations (3):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States
- Prof. Michael Blauth, Innsbruck, Tyrol, Austria
- Universitätsspital Basel, Basel, Basel, Switzerland